CLINICAL TRIAL: NCT05612776
Title: High Intensity Interval Training (HIIT) vs Heart Rate Variability (HRV) Training for Cardiac and Functional Rehabilitation After Stroke
Brief Title: HIIT vs HRV-based Training for Rehabilitation After Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad de Almeria (Other)
Collaborators: CEINSA, University of Almeria (Unknown)
Responsible Party: Principal Investigator, María Carrasco Poyatos, Principal Investigator, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AHIITATE
Record Dates: First submitted 2022-07-19; First posted 2022-11-10 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Stroke; Cardiac Disease; Ischemic Stroke; Ischemic Heart Disease; Stroke, Ischemic
Keywords: Heart Rate Variability; HIIT; cardiac rehabilitation; safety; adherence; VO2peak
MeSH Terms: conditions — Stroke; Heart Diseases; Ischemic Stroke; Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIIT-based training (Experimental): The HIIT group will train according to a predefined high intensity training program
  Interventions: Other: HIIT
- HRV-based training (Experimental): The training prescribed to the HRV group will depend on the subjects' diary HRV
  Interventions: Other: HRV

INTERVENTIONS:
Other: HIIT — HIIT training will consist of performing high intensity intervals along with passive rests. The intensity of the exercise will be progressively increased and the rest time will be decreased. All participants will perform the same training according to the maximum heart rate reached in the Bruce test.
  Arms: HIIT-based training
Other: HRV — The intervention group will perform HRV-based training, measuring HRV every day before training in order to obtain HRV normality ranges for each participant. If the HRV value is within the normal range, the participant will perform a high intensity training but if the HRV value is below the normal range, the participant will perform a continuous training at low intensity as active rest.
  Arms: HRV-based training

SUMMARY:
Consequences of stroke are manyfold but all of them are important factors on the long-term outcomes of rehabilitation, becoming an important health problem with requires health strategies with advanced age. High intensity interval training (HIIT) is an efficient training protocol used in cardiac rehabilitation programs, but owing to the inter-individual variability in physiological responses to training associated to cardiovascular diseases, the exercise dose received by each patient should be closely controlled and individualized to ensure the safety and efficiency of the exercise program. The heart rate variability (HRV) is actually being used for this purpose, as it is closely linked to de parasympathetic nervous system activation. In this way, higher scores in HRV are associated with a good cardiovascular adaptation. The objective of this protocol is to determine the effect of HIIT compared with HRV-guided training on cardiorespiratory fitness, heart rate variability, functional parameters, body composition, quality of life, inflammatory markers, cognitive function, and feasibility, safety and adherence in patients after stroke undertaking an 8-week cardiac rehabilitation program. This will be a cluster-randomized controlled protocol in which patients after stroke will be assigned to an HRV-based training group (HRV-G) or a HIIT-based training group (HIIT-G). HIIT-G will train according to a predefined training program. HRV-G training will depend on the patients' daily HRV. The peak oxygen uptake (VO2peak), endothelial and work parameters, the heart rate variability, the functional parameters, the relative weight and body fat distribution, the quality of life, the inflammatory markers, the cognitive function, and the exercise adherence, feasibility and safety will be considered as the outcomes. It is expected that this HRV-guided training protocol will improve functional performance in the patients after stroke, being more safe, feasible and generating more adherence than HIIT, providing a better strategy to optimize the cardiac rehabilitation interventions.

ELIGIBILITY:
Inclusion Criteria:

* left ejection fraction higher than 30% after stroke
* aged between 18 and 80 years old

Exclusion Criteria:

* presence of absolute or relative contraindications for accomplishing the treadmill test, indicated by the Spanish Society of Cardiology
* being treated for other diseases, or regularly taking a drug(s) that has a direct or indirect effect on the nervous system (e.g., anxiolytics, antidepressants or neuroleptics)
* absence of medication to control the cardiovascular disease or its modification during the intervention
* people who are participating or have participated in the previous three months in other similar exercise programs
* not performing at least 80% of the workouts during the intervention

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Peak oxygen uptake (VO2peak) changes | baseline and week 8
  According to the Spanish Society of Cardiology, the modified Bruce procotol will be used as a treadmill test, as it is indicated for people considered to be at high risk and the elderly.

SECONDARY OUTCOMES:
Heart rate variability | every day before starting the intervention
  HRV is proposed to be measured at rest, just before the training session, in a laying position and over a 60 second period. Smartphone application known as "HRV4Training" will be used.
Functional performance | Baseline and week 8
  To measure functional capacity, the Senior Fitness Test battery will be used such as the "Six Minutes Walk Test" Or "Timed Up and Go Tests", as it has been used in previous studies in which a program based on high-intensity training has been implemented with elderly people.
Body mass index (BMI) | Baseline and week 8
  Height will be measured using a measuring rod (Seca 213), and the body mass index (BMI) will be calculated according to the formula: BMI = kg/m2.
Quality of life MacNew | Baseline and week 8
  the MacNew QLMI post-myocardial infarction quality of life questionnaire will be administered. Consists of a 27-question questionnaire answered on a scale of 1 to 7, where 1 means "always" and 7 means "never".
Number of participants with abnormal laboratory test results | baseline and week 8
  The blood analysis will include the lipid profile, the detection and quantification of plasma insuline and its' resistance.
Waist-to-hip ratio | Baseline and week 8
  As body fat distribution can vary substantially, and having into account that abdominal adiposity has been associated with coronary heart disease, Waist-to-hip ratio will be measured according to International Society for the Advancement of Kinanthropometry Standards.
Waist-to-height ratio | Baseline and week 8
  In the same way, waist-to-height ratio will be also measured as a recent systematic reviews with meta-analysis have proposed it as a better predictor of cardiovascular risk factors.
Cognitive function, spatial memory recognition test | baseline and week 8
  the spatial memory recognition test (ASMRT), a simple virtual reality based task for specific population like older adults and with proved sensitivity to gender differences
Cognitive function, virtual version of the Walking Corsi test | baseline and week 8
  the virtual version of the Walking Corsi test (VR_WalCT) will be used to measure topographical memory, as proved its' equivalency regarding the real environment one
Cognitive function, Trail Making Test | baseline and week 8
  the Trail Making Test (TMT) will be used to detect neurological disease and neuropsychological impairment through the cognitive domains of processing speed, sequencing, mental flexibility and visual-motor skills.
Exercise Adherence | up to 8 weeks
  Adherence will be assessed by the number of sessions completed by the participants. At least, the 80% of the sessions should be achieved to consider a successful adherence.
Feasibility study | up to 8 weeks
  Feasibility study will be considered as the compliance to the exercise protocol, and will be registered as the percentage of participants that finished every training session.
Safety study | up to 8 weeks
  Safety study will be measured as the numbers of adverse events occurred during the training sessions. They will be registered as mild, moderate and severe. Moreover, their relation to the exercise session will also be taken into account.

CONTACTS AND LOCATIONS:
Locations (1):
- CITE III, Almería, Spain